CLINICAL TRIAL: NCT00339690
Title: Dust Mite Allergen Reduction Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 999905166; 05-E-N166
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-11-27

CONDITIONS: Allergy
Keywords: Asthma; Allergy; Intervention; Behaviors; Test-Kit; Dust Mites Allergen
MeSH Terms: conditions — Hypersensitivity; Asthma; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (1):
- Test Kit Homes (Experimental): Households assigned to use the in-home test kit.
  Interventions: Other: MITE-T-FASTtest kit

INTERVENTIONS:
Other: MITE-T-FASTtest kit — The primary objective of this randomized intervention trial is to determine if the use of an inhome test kit, as an adjunct to education, results in greater reductions in dust mite allergen levels than the use of educational materials alone.

SUMMARY:
This study will determine whether use of an in-home test kit results in decreased dust mite allergen levels in homes of children who are sensitive or allergic to dust mites. Dust mite allergens come from dust mites - microscopic spider-like animals that feed on house dust. Dust mites are common anywhere there is dust, such as in carpeting and beds. Some people are allergic to dust mite allergens and may develop asthma from living near them.

People who live in the Research Triangle Park area of North Carolina who have a child between 5 and 15 years old with a dust mite allergy or sensitivity may be eligible for this study. Participants must plan to remain in the same house for at least 12 months from the start of the study. At least half the floor of the child's room must be carpeted.

Participants are given materials on how to reduce dust mite allergens in their home. Study staff visit participants' homes three times over a 12-month period to ask questions about the home, home cleaning habits, and participants' experiences with home test kits (see below) for measuring dust mite allergen. At each visit, staff collect dust samples from the child's bedroom, the parents' bedroom, and the living room. The dust samples are analyzed in the laboratory for dust mite allergens and the results are given to the participants at the end of the study.

Participants are also given four home test kits for measuring dust mite allergen in the home. At the first home visit, staff instruct the participants on how to use the kits and answer any questions they may have. The kits are mailed at certain times during the study for the participants to use to measure allergen and send the results to the study investigators in a pre-paid addressed envelope.

A control group is given educational materials but no test kits.

DETAILED DESCRIPTION:
Sensitization to dust mite allergens is a major risk factor for the development and exacerbation of asthma. Asthmatics and others with dust mite allergies often implement strategies to avoid dust mite exposure, but lack objective evidence that their efforts are successful in reducing dust mite populations. Recently developed in-home test kits have introduced the capability to monitor the effectiveness of allergen reduction strategies by providing an affordable, simple way to measure dust mite allergens on a regular basis. The primary objective of this study is to determine if use of an in-home test kit result in decreased dust mite allergen levels in homes of children sensitive or allergic to dust mites. A secondary objective is to determine if use of an in-home test kit result in attitudinal and/or behavioral changes related to implementing and maintaining dust mite reduction strategies.

This study is a randomized controlled intervention trial designed to test the efficacy of an in-home test kit in influencing behaviors to reduce dust mite allergen levels. Households will be recruited through flyers and screened for eligibility through a recruitment call line. Study participants will be randomly assigned to a treatment or control group. The treatment group will receive educational materials and an in-home test kit at set intervals, while the control group will receive educational materials alone.

Vacuumed dust samples will be collected and delivered to the NIEHS laboratory for ELISA-based measurements of the dust mite allergens Der f 2 and Der p 2. A questionnaire will be used to collect information on home characteristics and on dust mite reduction attitudes and behaviors. The Precaution Adoption Process Model (PAPM) will be used to assess changes in attitudes and behaviors. Data will be collected at baseline, 6-months, and 12-months.

The primary statistical analysis will measure the change in allergen concentrations from baseline to month 12. This change will be compared between the two study arms using a generalized linear model to test the null hypothesis of no difference between groups. In secondary analyses, data from each sampling location will be analyzed separately and changes from 0-to-6 and 6-to-12 months will be compared between the treatment and control groups. Data from the questionnaire and baseline home visits will be analyzed for each group to determine PAPM stages and transitions. The results from this study will be used by NIEHS to plan future primary and secondary asthma prevention trials.

ELIGIBILITY:
* INCLUSION CRITERIA:

Live in Triangle area.

Plan to remain in the same house for at least 12 months.

Child in household aged 5 to 15 with allergy or sensitivity to dust mites (self-reported by parent or guardian, and a doctor's diagnosis of dust mite allergy or sensitivity is not required, i.e., if the parent or guardian believes or suspects that the child is allergic or sensitive to dust mites, that is sufficient).

Child sleeps in own bed at least 3 nights a week.

Child's room has carpeting on at least 50% of the floor.

Parents do not currently have dust mite protective mattress covers on the bed.

At least one of the two bedroom surfaces must have Group 2 dust mite allergen levels of greater than or equal to 2 microliter/g with the ELISA test AND greater than or equal to 2 microliter/g on at least one of the two Mite-T-Fast tests for inclusion.

EXCLUSION CRITERIA:

Does not meet inclusion criteria.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2005-06-06; Primary Completion 2009-02-11 (Actual); Study Completion 2009-02-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in the log-transformed (Der f 2 + Der p 2) allergen concentrations for the child s bed and bedroom floor. | Baseline, and months 6 and 12
Data from each of the six sampled locations (child s bed, child s bedroom floor, living room floor, parent s bed, and parent s floor) are analyzed separately, and changes are compared between the treatment and control groups. | Baseline, and months 6 and 12

SECONDARY OUTCOMES:
Data from the questionnaire and observation form will be used toaddress the secondary study objective to determine if use of an in-home test kit results in a change in dust mite reduction attitudes and behaviors. | Baseline, and months 1, 2, 5, 6, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C Zeldin, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Constella Group, Inc., Durham, North Carolina, United States

REFERENCES:
- [Background] Weiss KB, Sullivan SD. The health economics of asthma and rhinitis. I. Assessing the economic impact. J Allergy Clin Immunol. 2001 Jan;107(1):3-8. doi: 10.1067/mai.2001.112262. PMID 11149982
- [Background] Gergen PJ, Turkeltaub PC. The association of individual allergen reactivity with respiratory disease in a national sample: data from the second National Health and Nutrition Examination Survey, 1976-80 (NHANES II). J Allergy Clin Immunol. 1992 Oct;90(4 Pt 1):579-88. doi: 10.1016/0091-6749(92)90130-t. PMID 1401641
- [Background] Platts-Mills TA, Vervloet D, Thomas WR, Aalberse RC, Chapman MD. Indoor allergens and asthma: report of the Third International Workshop. J Allergy Clin Immunol. 1997 Dec;100(6 Pt 1):S2-24. doi: 10.1016/s0091-6749(97)70292-6. No abstract available. PMID 9438476
- [Derived] Winn AK, Salo PM, Klein C, Sever ML, Harris SF, Johndrow D, Crockett PW, Cohn RD, Zeldin DC. Efficacy of an in-home test kit in reducing dust mite allergen levels: results of a randomized controlled pilot study. J Asthma. 2016;53(2):133-8. doi: 10.3109/02770903.2015.1072721. Epub 2015 Aug 24. PMID 26308287